CLINICAL TRIAL: NCT01413841
Title: Phase II Randomised Study of Nasal Oxygen Treatment for Pain Relief During Percutaneous Coronary Interventions
Brief Title: Effect of Oxygen During Percutaneous Coronary Intervention for Pain Relief
Acronym: OXYPAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DELUCA2
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Angina
Keywords: PCI; oxygen
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal oxygen (Active Comparator): 3 liter per minute
  Interventions: Drug: Nasal oxygen
- Nasal Air (Placebo Comparator): 3 l regular nasal air
  Interventions: Drug: Regular nasal air

INTERVENTIONS:
Drug: Nasal oxygen — 3 l oxygen
  Arms: Nasal oxygen
Drug: Regular nasal air — 3 l nasal air
  Arms: Nasal Air

SUMMARY:
Nasal oxygen is widely used as pain relief against ischemic pain during Percutaneous Coronary Intervention (PCI). However, to our knowledge no randomised clinical trials have tested this. In contrast, oxygen causes coronary artery vasoconstriction in man. Furthermore, a recent Cochrane meta-analysis has shown no evidence of beneficial effect of oxygen for patients with acute myocardial infarction (with normal blood saturation. The investigators therefore wanted to examine if oxygen reduces ischemic pain during PCI for stable angina or NSTEMI.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina or NST-ACS undergoing PCI

Exclusion Criteria:

* Blood oxygen <95%
* Cognitive dysfunction
* STEMI
* Intubation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Chest pain measured with VAS | 1 h
  After PCI patient is asked in a double blinded about maximum chest during PCI.

SECONDARY OUTCOMES:
Troponin-levels after PCI | 2 days
  Peak troponin the first days after PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Skane University Hospital, Lund, Lund, Sweden

REFERENCES:
- [Derived] Zughaft D, Bhiladvala P, Van Dijkman A, Harnek J, Madsen Hardig B, Bjork J, Ekelund U, Erlinge D. The analgesic effect of oxygen during percutaneous coronary intervention (the OXYPAIN Trial). Acute Card Care. 2013 Sep;15(3):63-8. doi: 10.3109/17482941.2013.822083. PMID 23957447